CLINICAL TRIAL: NCT03503877
Title: Aneuploidy Rates and Morphokinetic Parameters in Sibling Embryos Cultured in Distinct Culture Media
Brief Title: Media, Morphokinetics, and Mosaicism
Acronym: 3M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-22331
Record Dates: First submitted 2018-02-07; First posted 2018-04-20 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Embryonic Mosaicism; Embryo Culture Media; Embryo Morphokinetics; Infertility
MeSH Terms: conditions — Infertility | interventions — Fetoscopes

STUDY DESIGN:
Intervention Model Description: sibling embryo study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SAGE Media (Other): SAGE single-step MEDIA
  Interventions: Device: EmbryoScope Plus; Other: SAGE MEDIA
- GLOBAL Media (Other): LIFE GLOBAL single-step MEDIA
  Interventions: Device: EmbryoScope Plus; Other: GLOBAL MEDIA

INTERVENTIONS:
Device: EmbryoScope Plus — All embryos will be cultured in the EmbryoScope Plus to obtain morphokinetic data
Other: GLOBAL MEDIA — Embryos will be cultured in GLOBAL media
  Arms: GLOBAL Media
Other: SAGE MEDIA — Embryos will be cultured in SAGE media
  Arms: SAGE Media

SUMMARY:
Embryonic aneuploidy is the underlying etiology for the majority of failed implantation and miscarriage. Preimplantation genetic screening (PGS) with transfer of a euploid embryo has been advocated as a strategy for increasing live birth rates with a single embryo transfer. Culturing embryos to the blastocyst stage for trophectoderm biopsy is a requirement for PGS. Several commercially-available single-step embryonic culture media with varying composition have been established for use in the IVF laboratory. Early reports have suggested differences in clinical outcomes, such as aneuploidy and miscarriage rates, with distinct culture media currently in standard use. However, there have been no clinical trials demonstrating the superiority of any one commercially-available culture media formulation. As a result, clinics use media with varying composition based upon familiarity and cost.

ELIGIBILITY:
Inclusion Criteria:

All subjects planning blastocyst culture for preimplantation genetic screening (PGS) will be offered enrollment.

Antral Follicle Count (AFC) >8 Male and female partner > 18 years of age

Exclusion Criteria:

Female partner age >42 years of age Cleavage stage biopsy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Rosen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between February 2018 and November 2019. All individuals planning in vitro fertilization with intent for blastocyst culture and PGT-A at UCSF Center for Reproductive Health were offered enrollment prior to their treatment cycle
Pre-assignment Details: Of 200 subjects enrolled, 1 subject was pregnant before her planned IVF cycle, 8 subjects were canceled prior to retrieval, 3 chose to withdraw from the study, 11 were found to be ineligible and 1 was withdrawn by study personnel due to the conversion to an oocyte cryopreservation cycle. As a result, 176 subjects underwent egg retrieval. Of these, 49 were removed from analysis for not having paired embryos and 127 had paired embryo sets in each culture arm and were able to complete the study.
Units Other Than Participants: Paired embryo sets
Period: Overall Study
Arm/Group | SAGE Media | GLOBAL Media
Started | 127; 127 Paired embryo sets | 127; 127 Paired embryo sets
Completed | 127; 127 Paired embryo sets | 127; 127 Paired embryo sets
Not Completed | 0; 0 Paired embryo sets | 0; 0 Paired embryo sets

BASELINE CHARACTERISTICS:
Units Other Than Participants: Paired embryo sets
Groups:
- All Study Participants: All study participants had paired embryo sets in each culture arm (SAGE Media or GLOBAL Media).
Arm/Group | All Study Participants
Number analyzed (Participants) | 127
Number analyzed (Paired embryo sets) | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 127
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 127

OUTCOME MEASURES:

1. Primary Outcome: Aneuploidy Rates
Description: number of embryos with abnormal chromosome number over total number of embryos biopsied (%)
Time Frame: Preimplantation Genetic Testing at blastocyst stage of embryo development, 2 weeks from start of IVF treatment
Measure: Mean (Standard Deviation); unit: percentage of embryos
Units Other Than Participants: Paired embryo sets
Arm/Group | SAGE Media | GLOBAL Media
Number analyzed (Participants) | 127 | 127
Number analyzed (Paired embryo sets) | 127 | 127
percentage of embryos | 56.1 (34.4) | 62.3 (34)
Statistical Analysis 1: Comparison: SAGE Media vs GLOBAL Media; Test type: Superiority; p = 0.07, Wilcoxon signed-rank testing

2. Secondary Outcome: Embryo Quality
Description: Fraction of freezable quality embryos (6 cells or greater, grades 1-2 for symmetry and fragmentation), (%).
Time Frame: 2 weeks from start of IVF treatment
Measure: Mean (Standard Deviation); unit: percentage of embryos
Units Other Than Participants: Paired embryo sets
Groups:
- Sage Media: SAGE single-step MEDIA EmbryoScope Plus: All embryos will be cultured in the EmbryoScope Plus to obtain morphokinetic data SAGE MEDIA: Embryos will be cultured in SAGE media
- Global Media: LIFE GLOBAL single-step MEDIA EmbryoScope Plus: All embryos will be cultured in the EmbryoScope Plus to obtain morphokinetic data GLOBAL MEDIA: Embryos will be cultured in GLOBAL media
Arm/Group | Sage Media | Global Media
Number analyzed (Participants) | 127 | 127
Number analyzed (Paired embryo sets) | 127 | 127
percentage of embryos | 45.7 (31.1) | 45.6 (30.8)
Statistical Analysis 1: Comparison: Sage Media vs Global Media; Test type: Superiority; p = 0.89, Wilcoxon signed-rank testing

3. Secondary Outcome: Embryonic Mosaicism
Description: Fraction of embryos given mosaic diagnosis. Embryonic mosaicism is defined as having partial aneuploidy (20-80% aneuploid). Low-level mosaicism is defined as 20-40% whereas high-level mosaicism is defined as 40-80%.
Time Frame: Preimplantation Genetic Testing at blastocyst stage of embryo development, 2 weeks from start of IVF treatment
Measure: Mean (Standard Deviation); unit: percentage of embryos
Units Other Than Participants: Paired embryo sets
Arm/Group | SAGE Media | GLOBAL Media
Number analyzed (Participants) | 127 | 127
Number analyzed (Paired embryo sets) | 127 | 127
percentage of embryos
  High Mosaic expression rate (40-80%) | 15.9 (25.7) | 18.9 (30.5)
  Low Mosaic expression rate (20-40%) | 1.0 (5.9) | 2.2 (9.0)
Statistical Analysis 1: Comparison: SAGE Media vs GLOBAL Media; Test type: Superiority; p = 0.54, Wilcoxon signed-rank testing — High mosaicism
Statistical Analysis 2: Comparison: SAGE Media vs GLOBAL Media; Test type: Superiority; p = .20, Wilcoxon signed-rank — Low mosaicism

4. Secondary Outcome: Embryo Morphokinetics
Description: time to first and all subsequent cell cleavages
Time Frame: 2 weeks from start of IVF treatment
Measure: Mean (Standard Deviation); unit: Hours
Units Other Than Participants: Paired embryo sets
Arm/Group | SAGE Media | GLOBAL Media
Number analyzed (Participants) | 127 | 127
Number analyzed (Paired embryo sets) | 127 | 127
Hours
  2 cell formation | 28.1 (3.9) | 28.4 (4.3)
  3 cell formation | 38.5 (6.6) | 39.5 (6.6)
  4 cell formation | 40.6 (5.3) | 41.2 (6)
  5 cell formation | 50.6 (6.5) | 52.3 (8.2)
  6 cell formation | 54.5 (8.3) | 55.4 (7.6)
  7 cell formation | 58.2 (8.1) | 58.8 (8.6)
  8 cell formation | 61.9 (8.7) | 62.5 (9)
  Morula Formation | 92 (8.9) | 93.4 (8.6)
  Start of Blastulation | 102.6 (8.1) | 104 (8.2)
  Blastocyst Formation | 110.6 (7.8) | 111.8 (7.6)
  Expanded Blastocyst Formation | 120.3 (8.1) | 122.5 (8.2)
Statistical Analysis 1: Comparison: SAGE Media vs GLOBAL Media; Test type: Superiority; p = 0.01, Wilcoxon signed-rank testing — Time to Expanded Blastocyst

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | SAGE Media | GLOBAL Media
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/127
Other Adverse Events (participants affected / at risk) | 0/127 | 0/127

LIMITATIONS AND CAVEATS:
A limitation of our study is the absence of long-term outcome data including pregnancy outcomes and offspring health data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03503877/Prot_SAP_000.pdf